CLINICAL TRIAL: NCT00001450
Title: Phase II Trial of a 96-Hour Continuous Infusion of Paclitaxel Followed by Cisplatin for Patients With Stage III/IV and Relapsed NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950198; 95-C-0198
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Neoplasms
Keywords: Chemotherapy; In Vitro Testing; Infusional; Lung Neoplasm; Pharmacokinetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Paclitaxel; Cisplatin

INTERVENTIONS:
Drug: paclitaxel
Drug: cisplatin

SUMMARY:
This is a Phase II study of paclitaxel (Taxol R) administered as a 96-hour (4 day) continuous infusion followed by a bolus of cisplatin for previously untreated patients with stage III/IV or relapsed non-small cell lung cancer (NSCLC). The goal of this phase II study is to determine the response rate of this infusional paclitaxel and bolus cisplatin regimen in patients with advanced NSCLC.

DETAILED DESCRIPTION:
This is a Phase II study of paclitaxel (Taxol R) administered as a 96-hour (4 day) continuous infusion followed by a bolus of cisplatin for previously untreated patients with stage III/IV or relapsed non-small cell lung cancer (NSCLC). The goal of this phase II study is to determine the response rate of this infusional paclitaxel and bolus cisplatin regimen in patients with advanced NSCLC. In addition, the plasma levels of paclitaxel will be measured, and the in vitro paclitaxel chemosensitivity of the tumor cells from as many patients as possible will be determined. This will allow further study of the relationship between in vitro drug sensitivity, achievable plasma concentrations of paclitaxel, and patients' response to therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically confirmed non-small cell lung cancer, including: Squamous cell carcinoma, Adenocarcinoma, Large cell carcinoma, Mixed histologies in the absence of a predominant small cell component.

Eligible Stages Include:

Stage IV, Stage IIIA/B ineligible for resection or radiotherapy, Postsurgical recurrence that is histologically or cytologically proven.

CNS Metastases Allowed Provided:

Radiotherapy completed prior to entry.

No requirement for concurrent steroids.

No carcinomatous meningitis.

No epidural metastases.

Measurable disease not required.

PRIOR/CONCURRENT THERAPY:

Biologic Therapy: Not specified.

Chemotherapy: No prior chemotherapy for lung cancer.

Endocrine Therapy: Not specified.

Radiotherapy: No prior chest irradiation for lung cancer.

Surgery: Prior surgery allowed.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance Status: ECOG 0-2.

Hematopoietic:

Absolute granulocyte count greater than 2,000.

Platelet count greater than 100,000.

Hepatic: Bilirubin no greater than 1.5 mg/dL.

Renal: Creatinine no greater than 1.5 mg/dL.

Cardiovascular:

No CHF unless fully compensated.

No second- or third-degree heart block.

No uncontrolled, symptomatic atrial dysrhythmia except sinus bradycardia.

No sustained ventricular tachycardia.

No MI within 3 months.

OTHER:

No uncontrolled infection unless due to an obstructed bronchus.

No major psychiatric problems requiring hospitalization.

No psychotropic medications such as phenothiazines.

No contraindication to transfusion, if required.

No second malignancy within 5 years except: Nonmelanomatous skin cancer.

In situ cervical cancer.

No pregnant or nursing women.

Effective contraception required of fertile patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58
Dates: Start 1995-09; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States